CLINICAL TRIAL: NCT02421874
Title: Development, Usability Testing, and Effectiveness Evaluation of Wraparound Team Monitoring System
Brief Title: Development and Testing of an Electronic Behavioral Health Record Specific to the Wraparound Care Coordination Process
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Eric Bruns, Associate Professor, Psychiatry, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2R42MH095516 (NIH)
Record Dates: First submitted 2015-04-10; First posted 2015-04-21 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Serious Emotional Disturbance of Youth
Keywords: Patient care team; Care management; Electronic health records

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Use of electronic health record / outcomes monitoring (Experimental): Use of electronic health record / outcomes monitoring via a specified electronic behavioral health information system
  Interventions: Behavioral: Wraparound Team Monitoring System electronic health record
- education about outcomes monitoring (Active Comparator): Care coordination as usual with education about fidelity and outcomes monitoring but no use of EBHIS
  Interventions: Behavioral: Education about fidelity maintenance and monitoring

INTERVENTIONS:
Behavioral: Wraparound Team Monitoring System electronic health record — Wraparound Team Monitoring System (Wrap-TMS) is a web-based, electronic behavioral health information system (EBHIS) for the most widely implemented care coordination model in children's behavioral health, the wraparound process
  Arms: Use of electronic health record / outcomes monitoring
Behavioral: Education about fidelity maintenance and monitoring — As an active comparator, we will educate practitioners randomized to the control condition about the importance of maintaining fidelity and monitoring fidelity and progress via a 3 hour training.
  Arms: education about outcomes monitoring

SUMMARY:
The purpose of this Phase II Small Business Technology Transfer (STTR) project is to complete development and evaluate usability and effectiveness of the Wraparound Team Monitoring System (Wrap-TMS), a web-based, electronic behavioral health information system (EBHIS) for the most widely implemented care coordination model in children's behavioral health, the wraparound process. Though wraparound is now considered "evidence-based," implementation in the real world often fails to conform to standards of fidelity and/or use objective data to guide management, supervision, and clinical decision making. Availability of such a system will support efficiency, implementation quality and fidelity, and outcomes for youths enrolled in wraparound. Wrap-TMS features functionality for data entry, management, and basic reporting for the full array of data and information elements needed to manage an integrated care coordination initiative for youths with serious emotional and behavioral disorder (SEBD). In light of our success in Phase I, subsequent partnerships with federal agencies, and inquiries of interest from several states and over 20 provider and managed care organizations, in this Phase II STTR the investigators will complete development of Wrap-TMS, followed by a randomized controlled effectiveness study comparing n=25 wraparound facilitators who use Wrap-TMS serving n=100 families to 25 non-user facilitators serving 100 families on practitioner, implementation, and youth/family outcomes. The evaluation will test two primary hypotheses:

1. Compared to facilitators in the control group, wraparound facilitators trained to use Wrap-TMS will demonstrate (a) greater use of data and feedback in service delivery; (b) greater fidelity to the wraparound process; (c) higher self-reported teamwork, working alliance, and satisfaction with the intervention; and (d) more positive attitudes toward standardized assessment.
2. Compared to the control group, parents of youths receiving services from facilitators trained to use TMS will report (a) greater goal clarity, (b) more data collection and use (c) greater satisfaction with services and progress, (d) better fidelity to wraparound, (e) more effective team functioning, (f) greater treatment alliance, and (f) better youth outcomes including greater progress and improved symptoms and functioning.

ELIGIBILITY:
Inclusion Criteria:

* Parent or legal guardian of a youth aged 6-17 with SEBD (serious emotional and behavioral disorder): at least one MH (mental health) diagnosis that results in long-term (>6 mos) impairment in home, school and/or community functioning).

Exclusion Criteria:

* Non English speaking parents
* Foster parents

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2015-07; Primary Completion 2016-11 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
more effective teamwork (Team Climate Inventory (TCI) | 6 months
  Team Climate Inventory (TCI). The TCI is a 38-item survey that evaluates five relevant aspects of health care teamwork (Shared Vision, Participation safety, Support for Innovation, Task orientation, Interaction frequency) using a 5 point Likert scale. Assessed at 4 mos. post enrollment
treatment alliance (Working Alliance Inventory (WAI) | 6 months
  Working Alliance Inventory (WAI) is a widely used rating scale designed to measure the working alliance between counselors and clients. Assessed at 4 mos. post enrollment
improved youth functioning (Top Problem Assessment (TPA) | 6 months
  Top Problem Assessment (TPA) is a consumer-focused index the severity of the top three problems nominated by the parent, on a scale of 0-10. Assessed at BL, 1, 2, 3, 4 mos.

SECONDARY OUTCOMES:
parent and provider satisfaction (Parent and Child Satisfaction Scales) | 3 months
  Parent and Child Satisfaction Scales reliably measure five dimensions of satisfaction, each with 1 Likert scale item, including: (1) access and convenience, (2) child's treatment process and relationship with providers, (3) parent and family services, satisfaction with progress, and (5) global satisfaction. Assessed at 4 mos post enrollment
attitudes toward standardized assessment (Attitudes toward Standardized Assessment Scale (ASA)105) | 3 months
  Attitudes toward Standardized Assessment Scale (ASA)105. A 22-item measure of clinician perceptions and attitudes about using standardized assessments in their clinical practice. Items are scored on a 1 (Strongly Disagree) to 5 (Strongly Agree) scale and yield 3 subscales with adequate or better reliabilities: Benefit over Clinical Judgment, Psychometric Quality, and Practicality. Administered to practitioners at baseline and 4 mos.

CONTACTS AND LOCATIONS:
Overall Officials: Eric J Bruns, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bruns EJ, Hook AN, Parker EM, Esposito I, Sather A, Parigoris RM, Lyon AR, Hyde KL. Impact of a Web-Based Electronic Health Record on Behavioral Health Service Delivery for Children and Adolescents: Randomized Controlled Trial. J Med Internet Res. 2018 Jun 14;20(6):e10197. doi: 10.2196/10197. PMID 29903701